CLINICAL TRIAL: NCT06796114
Title: Identification of Innovative Biomarkers to Predict Outcomes in Hepatocellular Carcinoma Treated With Tremelimumab and Durvalumab
Acronym: PREDICT-HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-931; 2024-A02783-44 (Other: IDRCB)
Record Dates: First submitted 2025-01-10; First posted 2025-01-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: biomarker, immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood sample (Experimental)
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — A total of 48 ml of blood will be collected at baseline (before STRIDE initiation):
  * 6 EDTA 6 ml tubes for PBMC collection
  * 2 EDTA 6 ml tube for plasma collection

SUMMARY:
Several cancer immunotherapies that target the PD-L1/PD-1 pathway (i.e., checkpoint inhibitors) show promising clinical activity in patients with HCC. In particular, atezolizumab selectively targets PD-L1 to prevent interaction with receptors PD-1 and B7-1, thus reversing T-cell suppression. Moreover, atezolizumab in combination with bevacizumab, a monoclonal antibody that targets VEGF and inhibits angiogenesis, is associated with an objective response rate of 27.3% (Cheng et al. 2021; Finn et al. 2020). This tumor response has led to FDA (Food and Drug Administration) and EMA (European Medicines Agency) approvals, in first-line treatment in unresectable HCC.

Combinations studies evaluating anti-CTLA4 and anti-PD1/PDL1 antibodies displayed greater benefits (Abou-Alfa et al. 2022). In the Phase 3 HIMALAYA study (NCT03298451) in uHCC, a single priming dose of tremelimumab (anti-CTLA-4) plus durvalumab (anti-PD-L1) in the STRIDE (Single Tremelimumab Regular Interval Durvalumab) regimen significantly improved OS versus sorafenib; durvalumab monotherapy was noninferior to sorafenib for OS.

In the HIMALAYA study, STRIDE regimen induced long term survival (defined as the absence of progression above 36 months following inclusion) in 103 out of the 393 patients exposed to this strategy (26%).

The identification of biomarkers allowing the prediction of immunotherapy efficacy in HCC is still an unmet medical need.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Histologically confirmed hepatocellular carcinoma
3. Locally advanced, metastatic, or unresectable disease
4. Patient who had not previously received systemic anti-cancer treatment and are eligible to STRIDE therapy according to investigator decision in routine care and who have no contraindications to STRIDE treatment according to approved product label.
5. Measurable disease defined according to RECIST v1.1 guidelines (Note: Previously irradiated lesions can be considered as measurable disease only if disease progression has been unequivocally documented at that site since radiation.)
6. Age ≥ 18 years
7. Patient affiliated to or beneficiary of French social security system
8. Ability to comply with the study protocol, in the Investigator's judgment.

Exclusion Criteria:

1. Patients previously exposed to anti-tumor immunotherapy as anti-PD-1, anti-PD-L1, or anti-CTLA4 agent or any immune therapy.
2. Patient with any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study
3. Patient under guardianship, curatorship or under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-06-25 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
real-word overall survival | through study completion, up to a maximum of 24 months after the inclusion of the last patient
  defined as the delay from the date of treatment initiation to death from any cause

SECONDARY OUTCOMES:
real-word progression-free-survival | through study completion, up to a maximum of 24 months after the inclusion of the last patient
  defined as the delay from the date of treatment initiation to the disease progression or death from any cause whichever occurs first, evaluated by RECIST criteria v1.1 and mRECIST.
Objective Response Rate (ORR) | through study completion, up to a maximum of 24 months after the inclusion of the last patient
  defined as the addition of complete response and partial response rates, evaluated by RECIST citeria v1.1 and mRECIST
Disease control rate (DCR) | through study completion, up to a maximum of 24 months after the inclusion of the last patient
  defined as the addition of complete response, partial response, and stable disease rates evaluated by RECIST criteria v1.1 and mRECIST.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU de Besançon, Besançon
  - CH de Chalon sur Saône, Chalon-sur-Saône
  - CHU Grenoble, Grenoble
  - CH de Mulhouse, Mulhouse
  - Hôpital Beaujon - APHP, Paris
  - Hôpital Henri Mondor - APHP, Paris
  - Hôpital La Pitié Salpêtrière - APHP, Paris
  - ICANS, Strasbourg

IPD SHARING:
Plan to Share IPD: No